CLINICAL TRIAL: NCT05564598
Title: A Phase II Open-Label Randomized Study of Anti-Viral Antibiotic Therapy With and Without Familial (Maternal) Cytomegalovirus (CMV) Cytotoxic T Lymphocytes (CTLs) in Neonates With Moderate/Severe Maternal Acquired CMV Infection
Brief Title: CMV CTLs in Neonates With CMV Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 597; 1R01FD007837-01 (FDA)
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Congenital Cytomegaloviral (CMV) Disease
MeSH Terms: conditions — Disease | interventions — Valganciclovir; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 Safety Run-in (Experimental): The first 3 patients enrolled will receive both anti-viral medication and CMV CTLs, and treatment will be staggered every 28 days from the last dose of CMV CTLs from the prior patient.
  Interventions: Biological: CMV Cytotoxic T-Lymphocytes; Drug: Anti-viral Therapy
- Cohort 2 Antiviral medication + CMV CTLs (Experimental): Patients will receive both anti-viral medication and CMV CTLs
  Interventions: Biological: CMV Cytotoxic T-Lymphocytes; Drug: Anti-viral Therapy
- Cohort 2 Antiviral medication only (Active Comparator): Patients will only receive anti-viral therapy
  Interventions: Drug: Anti-viral Therapy

INTERVENTIONS:
Biological: CMV Cytotoxic T-Lymphocytes — Patients will receive maternal CMV CTLs on day 0. Additional doses of CMV CTLs may be re-infused at a minimum of every two weeks for a maximum of five total infusions (maximum 2.5 x 104 CD3/kg) only in patients not achieving a CR and no prior dose limiting toxicity of any prior dose.
  Other Names: CTLs
  Arms: Cohort 1 Safety Run-in; Cohort 2 Antiviral medication + CMV CTLs
Drug: Anti-viral Therapy — All patients will receive anti-viral therapy with one of the following:
  4.2.2 Valganciclovir Dosing: 16 mg/kg/dose PO q12h OR 4.2.3 Ganciclovir Dosing: 6 mg/kg/dose IV q12h
  Dose adjustments:
  * Reduce dose by 50% for ANC less than 500 cells/mm3
  * Hold the dose if ≤ 200 cells/mm3 until recovery ≥ 500 cells/mm3
  * Treatment will continue for 6 months
  Other Names: valganciclovir, ganciclovir

SUMMARY:
Patients with moderate or severe CMV disease less than 21 days old who have a maternal donor who has a CMV response to the peptivators will be screened.

All patients will receive treatment with valganciclovir or ganciclovir. There is a safety run in with treatment with CMV CTLs in cohort 1 and if found to be safe, will proceed to cohort 2 for randomization to receive antiviral therapy with or without CMV CTLs.

Funding source: FDA OOPD

DETAILED DESCRIPTION:
Given the vulnerability and poor outcomes of preterm neonates and neonates in general to viral infection, including the need for prolonged antiviral therapy for 6 or more months to achieve just modest improvements in sensorineural functions, CMV CTL therapy offers a promising alternative. CMV CTL treatment will build on the hosts innate immune capacity to create a more effective and permanent defense against collateral injury arising from CMV infections.

Patients who meet all inclusion/exclusion criteria with a maternal donor who meet all donor criteria will be enrolled onto study.

Cohort 1 is a safety run-in; the first 3 patients enrolled will be treated with anti-viral and CMV CTLs. The external DSMB will review the data from the first patient, and if there are no adverse events or dose-limiting toxicities observed, approve patient 2, and then 3, 28 days after the prior patients last CTL infusion. Assuming there are no adverse events in any of the first 3 patients, the study will proceed to Cohort 2.

Cohort 2 will be randomized 1:1 to either anti-viral treatment alone or anti-viral treatment plus CMV CTLs.

Patients who are randomized to receive CMV CTLs will get their first infusion on Day 0. If the patient fails to achieve a CR, they may receive one infusion every 2 weeks up to 5 maximum CMV CTL infusions as long as there are no DLTs or AEs observed

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤ 21 days of life
* Birth Weight: ≥ 2500 gms
* Gestational age: ≥ 34 weeks of age
* Diagnosis of CMV viremia, viruria, and/or infection:Either one or more:

Elevated CMV by RT-PCR in urine, saliva, CSF, or plasma; and/or Positive urine culture for CMV

- Moderate or Severe CMV Disease

Any one or more of the following attributable to congenital CMV infection:

* Thrombocytopenia (≤ 50,000 mm3)
* Multiple petechiae
* Hepatomegaly
* Splenomegaly
* Intrauterine growth retardation
* Increased transaminases
* Increased bilirubin
* Microcephaly
* Ventriculomegaly
* Intracerebral calcifications
* Periventricular echogenicity
* Cortical or cerebral malformation
* Chorioretinitis
* Severe neonatal hearing loss
* CMV DNA by PCR in CNS
* Increased WBC for age in CNS

  * Minimal Organ Criteria Hematological: ANC ≥ 750/mm3, HgB ≥ 8gm/dl, Platelets ≥ 20,000/kmm3 Renal: Serum creatinine ≤ 1.0 mg/dl Hepatic: ALT/SGOT ≤3x upper normal limits
  * Donor Availability: Maternal donor available with a T-cell response CMV MACS® PepTivators. the donor is considered suitable if the percentage of IFN-gamma+ T cells is > 0.01% after stimulation with PepTivators.

Exclusion Criteria -

* Patient receiving steroids (> 0.5 mg/kg prednisone equivalent) on the same day of CMV CTL infusion. Antenatal steroids for lung maturation will have been cleared prior to CMV diagnosis.
* Concomitant enrollment in another experimental clinical trial investigating the treatment of neonatal CMV viremia and/or infection.
* Any medical condition that could compromise participation in the study according to the investigator's assessment.
* Known history of HIV infection in the mother.
* Patient's legally authorized representative unwilling or unable to comply with the protocol or unable to give informed consent.

Ages: 0 Days to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of giving CMV CTLs combined with anti-viral therapy in neonates with CMV | 12 weeks
  the incidence and severity of Grade I-IV acute GVHD within 8 weeks that is probably or directly related to CMV-CTL infusion after last CMV CTL infusion will be evaluated to determine the safety profile of CMV CTLs in neonates
To determine response rates to treatment with CMV CTLS and anti-viral medication | 12 weeks
  response rates will be measured by monitoring CMV PCR levels. A complete response to CMV-CTLs will be those with undetectable viral load by qRT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Washington University, St Louis, Missouri
  - New York Medical College, Vallhala, New York
  - Nationwide Children's Hosptial, Columbus, Ohio